CLINICAL TRIAL: NCT02785809
Title: Recovery of Ovarian Function and Reserve Parameters After Discontinuation of Long-term Use of Oral Contraception: Is the Recovery Period Related to AMH?
Brief Title: Ovarian Function and Reserve Parameters After Discontinuation of Long-term Use of Oral Contraception
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anders Nyboe Andersen (Other)
Collaborators: Hvidovre University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Anders Nyboe Andersen, Professor M.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-16021266
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Oral Contraceptives; Long-term Use; AMH; Ovarian Reserve Parameters
Keywords: Oral contraceptives; long-term use; AMH; Ovarian reserve parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Withdrawal of bloodsamples (6 within a three months period) for analyses of reproductive hormones.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pausing oral contraceptive

SUMMARY:
The aim of this study is to investigate whether there is a correlation between anti-Müllerian hormone during long-term use of combined oral contraceptives and the recovery time before recovered menstrual cycle after discontinuation of oral contraceptives.

DETAILED DESCRIPTION:
Background:

Hormonal contraception is widely used among women worldwide; 50-89% of all women in the Western countries use oral contraception at some point in their lives. Oral contraceptives (OC) suppress the hypothalamic-pituitary-ovarian axis through a negative feedback of ethinyl estradiol and progestins and thereby potentially influence the markers of ovarian reserve due to a suppressed release of gonadotropins, which will impair the growth of antral follicles.

Methods and Materials:

Participants for this studies will be included through the Fertility Assessment and Counseling Clinic, Rigshospitalet, Herlev- and Hvidovre Hospital.

Inclusion criteria: Use of oral contraception (for study 3 at least during the last three years).

Exclusion criteria: Known infertility, known thyroid disease.

Aims:

Study 3: Investigate the ovarian reserve markers after discontinuation of OC over a period of three months in women with a history of long-term OC use. The women will be followed with serial ultrasounds and blood samples and will complete a menstrual calendar.

ELIGIBILITY:
Inclusion Criteria:

* Minimum three years of oral contraceptives.

Exclusion Criteria:

* Known infertility, known thyroid disease.

Ages: 26 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with a history of long term use of combine oral contraception for at least 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-05 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Time for recovered menstrual cycle after discontinuation of oral contraception | 6 months after discontinuation
Ovarian reserve parameters before and after discontinuation of combined oral contraception | 3 months after discontinuation

SECONDARY OUTCOMES:
Correlation between suppression of the pituitary gonodal axis during use of oral contraceptives and time for recovered menstrual cycle | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Selma K Landersoe, MD, Principal Investigator — Rigshospitalet, The Fertility Clinic
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, The Fertility Clinic, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alkema L, Chou D, Hogan D, Zhang S, Moller AB, Gemmill A, Fat DM, Boerma T, Temmerman M, Mathers C, Say L; United Nations Maternal Mortality Estimation Inter-Agency Group collaborators and technical advisory group. Global, regional, and national levels and trends in maternal mortality between 1990 and 2015, with scenario-based projections to 2030: a systematic analysis by the UN Maternal Mortality Estimation Inter-Agency Group. Lancet. 2016 Jan 30;387(10017):462-74. doi: 10.1016/S0140-6736(15)00838-7. Epub 2015 Nov 13. PMID 26584737
- [Background] van Heusden AM, Fauser BC. Residual ovarian activity during oral steroid contraception. Hum Reprod Update. 2002 Jul-Aug;8(4):345-58. doi: 10.1093/humupd/8.4.345. PMID 12206469
- [Derived] Landersoe SK, Larsen EC, Forman JL, Birch Petersen K, Kroman MS, Frederiksen H, Juul A, Nohr B, Lossl K, Nielsen HS, Nyboe Andersen A. Ovarian reserve markers and endocrine profile during oral contraception: Is there a link between the degree of ovarian suppression and AMH? Gynecol Endocrinol. 2020 Dec;36(12):1090-1095. doi: 10.1080/09513590.2020.1756250. Epub 2020 May 2. PMID 32362164